CLINICAL TRIAL: NCT02616809
Title: Effects of Standing and Light-intensity Activity on Ambulatory Blood Pressure and Blood Glucose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Noe Crespo, Assistant Professor, Arizona State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1306009298
Record Dates: First submitted 2015-11-24; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes; Hypertension; Sleep
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sitting (Experimental): Participants will sit continuously for 8 hours in a simulated office environment
  Interventions: Other: Maintaining posture and energy expenditure
- slow cycling (Experimental): Participants will cycle at regular hourly intervals during an 8-hr simulated office environment
  Interventions: Other: Increasing energy expenditure
- standing (Experimental): Participants will change posture (from sitting to standing) during hourly intervals for an 8-hr period in a simulated office environment
  Interventions: Other: Changing posture
- slow walking (Experimental): Participants will transition from sitting to slow walking on a treadmill desk at regular hourly intervals during an 8-hr period in a simulated office environment
  Interventions: Other: Increasing energy expenditure and changing posture

INTERVENTIONS:
Other: Maintaining posture and energy expenditure — Participants will sit continuously for 8-hrs during a simulated office environment
  Arms: Sitting
Other: Increasing energy expenditure — Participants will cycle slowly while seated in prescribed hourly intervals. This condition will increase energy expenditure while keeping a sitting posture
  Arms: slow cycling
Other: Changing posture — Participants will transition from sitting to standing in prescribed hourly intervals. This condition will change posture (sit to stand) while maintaining low energy expenditure
  Arms: standing
Other: Increasing energy expenditure and changing posture — Participants will transition from sitting to a walking workstation in prescribed hourly intervals. This condition will both increase energy expenditure and change posture.
  Arms: slow walking

SUMMARY:
This study aims to test the short-term effects of intermittent standing, slow cycling and slow walking, compared to sitting, on continuous blood glucose and ambulatory blood pressure among pre-hypertensive and pre-diabetic adults.

DETAILED DESCRIPTION:
This study will enroll 10 adults who will each complete four experimental conditions in random order. Each of the four experimental conditions are as follows: 1) sit continuously for 8 hours in a simulated office environment, 2) break-up sitting time with standing based on set hourly intervals, 3) break-up sitting time with slow-walking on a treadmill desk based on set hourly intervals, 4) increase energy expenditure by slow cycling based on set hourly intervals. Participants will completed each condition one week apart and dietary intake will be standardized by giving participants the same meals during each intervention condition. Study measures will include: anthropometrics (height and weight), blood pressure, fasting glucose, 24-continuous glucose monitoring, full-day ambulatory blood pressure monitoring, cognitive testing (cognitive performance), energy expenditure, physical activity via accelerometer, sleep via accelerometer, and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* pre-hypertensive (systolic blood pressure 120-139 mmHg, or diastolic blood pressure 80-89 mmHg)
* impaired fasting glucose (5.6-6.9 mmil/L)
* not meeting the physical activity guidelines for adults (>=150 min/wk of moderate-to-vigorous physical activity)

Exclusion Criteria:

* smoking, pregnancy, known coronary heart disease, orthopedic limitations for performing physical activity, taking medications to control high blood pressure or high blood glucose, special dietary requirements, and being advised by a doctor to avoid prolonged periods of sitting.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Evidence of change in blood pressure following changes in posture and increasing energy expenditure | single-day intervention
Evidence of change in blood glucose following changes in posture and increasing energy expenditure | single-day intervention